CLINICAL TRIAL: NCT01573104
Title: Evaluating the Utility of Urinary Proteomics and Novel Biomarkers in Acute Kidney Injury
Brief Title: Evaluating Novel Biomarkers in Acute Kidney Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Robert Docking (Other)
Responsible Party: Sponsor-Investigator, Dr Robert Docking, Clinical Research Fellow, University of Glasgow
Organization: University of Glasgow (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: RID-001
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Acute Kidney Injury
Keywords: Diagnosis; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury; Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biomarker group (Experimental): Patients undergoing CPB having proteomic assays, blood sampling and biomarker assays performed on D0, D1, D2 and D3
  Interventions: Other: Proteomic assay; Other: Blood sampling; Other: Biomarker sampling

INTERVENTIONS:
Other: Proteomic assay — Urine will be taken for proteomic assay at baseline, day 1 and day 2
Other: Blood sampling — Point of care testing of blood for NGAL/BNP at baseline, day 1 and day 2
Other: Biomarker sampling — Urine will be taken at baseline and day 1, day 2 for evaluation of renal biomarkers at later date

SUMMARY:
The investigators have a new technique of looking at urine to see whether it contains protein fragments that are released by damaged kidneys. These fragments seem to be more accurate than the current blood tests that the investigators use to diagnose renal failure. This technique needs to be validated with a group of patients that have a relatively high incidence of renal failure, cardiopulmonary bypass.

The investigators hypothesise that using novel markers of renal dysfunction will identify patients who go on to develop renal failure earlier, and in a higher number than the standard blood tests.

The investigators aim to collect urine from patients before going onto bypass, and then at Day 1 and Day 2 after bypass. This urine will be analysed for protein fragments, as well as other new markers of renal dysfunction. The investigators will also take blood at baseline and for the first two days in Cardiac Intensive Care, and compare the accuracy of the new tests with the 'gold standard' that is creatinine.

DETAILED DESCRIPTION:
The diagnosis of acute renal failure has been problematic, with a review showing 35 working definitions being used in the literature. This lack of clarity gave rise to the ADQI group creating the terminology of acute kidney injury (AKI). AKI has been used to give foundation to both the RIFLE and AKIN criteria, which have been shown to perform well in predicting critical care and hospital mortality. Their criteria are based on measuring increases of serum creatinine from baseline levels, and tallying this with weight-based urinary volumes. Problems with these techniques lie in having accurate baseline creatinine values, with the MDRD formula often proving inaccurate. Criticisms have also been levelled at using serum creatinine at all, given its variance with different body-mass compositions and fluid-balance status, as well as its relatively late rise in AKI compared to its utility in chronic renal failure.

Many novel biomarkers have been investigated in AKI, either serum or urine (cystatin-C, Il-18, KIM-1, NGAL). Results have been varied, with potential problems being lack of specificity to AKI, cost and the heterogeneous nature of patient populations in the various studies. NGAL has emerged as potentially the most specific to early AKI and additionally a number of commercially available assays are now available. Interest has been shown in the use of biomarker panels, allowing for improved sensitivity, albeit at a higher cost. Urinary proteomic analysis has been used as an investigative technique for AKI for the last ten years, but diverse populations and lack of blinding hampered early studies. A recent paper used techniques developed by collaborators on this proposal to improve the performance of proteomic assays, with impressive performance of these assays when looking at critically ill patients with AKI.

A problem with assessing the utility of diagnostic or screening tools for AKI in the critically ill is the heterogeneity of pathological insults, and the unpredictable early clinical course. This leads to difficulties in identifying control groups, and in capturing the evolution of AKI. We propose investigating the use of these novel biomarkers and proteomic techniques in the more homogenous group of patients undergoing cardiopulmonary bypass. This carries with it the benefits of thorough pre-operative testing with stable baseline measurements and a clearly definable renal insult in the form of bypass time. Post-bypass renal failure requiring RRT is estimated to occur in 1.5-2% of coronary artery grafting cases, and around 5% of combined graft/valve replacement cases; however, there is a far higher incidence of AKI as measured by creatinine rise and/or oliguria.

As part of standard operative technique patient's bladders are catheterised prior to the start of surgery and the first 100mls urine voided will be collected as the baseline sample. Venous blood will be taken at cannulation with serum spun and frozen for later analysis of NGAL (and any emergent biomarkers of AKI of interest). Finger prick blood sampling will be performed for baseline point of care analysis of NGAL/brain natriuretic peptide using the Alere platform.

Details of intra-operative conduct will be gathered from the computerised anaesthetic record and the cardiac perfusionist records including anaesthetic technique (volatile/TIVA), duration of bypass and perfusion pressures on bypass.

When in the Cardiac Intensive Care Unit (CICU) further 100mls urine will be collected at 24hrs after induction of anaesthesia, and at 48 hours. This will be a 'clean' sample (ie not from urine lying overnight). Accompanying laboratory values of serum creatinine will be collected for diagnosis of AKI and comparison to proteomic values. At the same point blood will be taken and stored for NGAL as well as finger prick measures using point of care NGAL/BNP.

Copies of the corresponding electronic ICU physiological records will be collated for data relating to cardiovascular parameters, diagnosis of AKI and use of vasopressors. APACHE-II scores will be calculated at 24 hours post admission in addition to daily SOFA scores. AKI will be defined as AKIN stage I (increase of serum creatinine >50% of baseline measurement, and/or urinary output <0.5ml/kg/hour for six hours) or RRT up to 48 hours post-surgery. Patient outcomes will be recorded in respect to CICU mortality, 90-day mortality, need for ongoing RRT, development of chronic kidney disease (moving from eGFR >60ml/min/1.73m2 pre-admission to eGFR <60ml/min/1.73m2 at hospital discharge).

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective cardiopulmonary bypass
* mental capacity
* able to understand written English

Exclusion Criteria:

* patient refusal
* surgical refusal
* chronic renal replacement therapy
* emergency procedures
* peri-operative use of ventricular assist devices
* pregnancy
* pre-operative exercise function NYHA IV
* severe chronic renal failure (eGFR <30ml/min/1.73m2).
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-11; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Development of acute kidney injury | Within two days of cardiopulmonary bypass
  Development of AKI will be defined by stage 1 of AKIN criteria (ie serum Creatinine >25% of baseline, or oliguria <0.5ml/kg/hr for 6 hours.

CONTACTS AND LOCATIONS:
Overall Officials: John Kinsella, MD, FRCA, Principal Investigator — University of Glasgow
Locations (1):
- Golden Jubilee National Hospital, Glasgow, United Kingdom